CLINICAL TRIAL: NCT03131895
Title: A Phase 1, Randomized, Open-Label, Single-Center, Single-Dose, Two-Period Two-Part Crossover Study in Healthy Subjects to Compare the Bioavailability of Dexlansoprazole From Dexlansoprazole Delayed-Release Capsules 30 mg and 60 mg Manufactured by Takeda GmbH Plant Oranienburg Relative to Dexlansoprazole Delayed-Release Capsules 30 mg and 60 mg Manufactured by Takeda Pharmaceutical Company Limited Osaka Plant
Brief Title: Bioequivalence Study of Dexlansoprazole Capsules From Two Manufacturing Plants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-390MR-1001; U1111-1184-2186 (Registry Identifier: WHO)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1, Sequence 1 (Regimen A, B) (Experimental): Dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (Regimen A [test]), orally, once on Day 1 of Period 1 following a 10 hour fast, followed by minimum of 5 day washout period, followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (Regimen B [reference]), orally, once on Day 1 of Period 2 following a 10-hour fast.
  Interventions: Drug: 30 mg dexlansoprazole capsules manufactured at TOB; Drug: 30 mg dexlansoprazole capsules manufactured at TPC
- Part 1, Sequence 2 (Regimen B, A) (Experimental): Dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (Regimen B [reference]), orally, once on Day 1 of Period 1 following a 10 hour fast, followed by minimum of 5 day washout period, followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (Regimen A [test]), orally, once on Day 1 of Period 2 following a 10-hour fast.
  Interventions: Drug: 30 mg dexlansoprazole capsules manufactured at TOB; Drug: 30 mg dexlansoprazole capsules manufactured at TPC
- Part 2, Sequence 3 (Regimen C, D) (Experimental): Dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (Regimen C [test]), orally, once on Day 1 of Period 1 following a 10 hour fast, followed by minimum of 5 day washout period, followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (Regimen D [reference]), orally, once on Day 1 of Period 2 following a 10-hour fast.
  Interventions: Drug: 60 mg dexlansoprazole capsules manufactured at TOB; Drug: 60 mg dexlansoprazole capsules manufactured at TPC
- Part 2, Sequence 4 (Regimen D, C) (Experimental): Dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (Regimen D [reference]), orally, once on Day 1 of Period 1 following a 10 hour fast, followed by minimum of 5 day washout period, followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (Regiment C [test]), orally, once on Day 1 of Period 2 following a 10-hour fast.
  Interventions: Drug: 60 mg dexlansoprazole capsules manufactured at TOB; Drug: 60 mg dexlansoprazole capsules manufactured at TPC

INTERVENTIONS:
Drug: 30 mg dexlansoprazole capsules manufactured at TOB — Dexlansoprazole delayed-release.
  Arms: Part 1, Sequence 1 (Regimen A, B); Part 1, Sequence 2 (Regimen B, A)
Drug: 30 mg dexlansoprazole capsules manufactured at TPC — Dexlansoprazole delayed-release.
  Arms: Part 1, Sequence 1 (Regimen A, B); Part 1, Sequence 2 (Regimen B, A)
Drug: 60 mg dexlansoprazole capsules manufactured at TOB — Dexlansoprazole delayed-release.
  Arms: Part 2, Sequence 3 (Regimen C, D); Part 2, Sequence 4 (Regimen D, C)
Drug: 60 mg dexlansoprazole capsules manufactured at TPC — Dexlansoprazole delayed-release.
  Arms: Part 2, Sequence 3 (Regimen C, D); Part 2, Sequence 4 (Regimen D, C)

SUMMARY:
The purpose of this study is to assess the bioavailability of dexlansoprazole from a 30 milligram (mg) or 60 mg delayed-release capsule manufactured at Takeda GmbH Plant Oranienburg, Germany (TOB) relative to that of dexlansoprazole from a 30 mg or 60 mg capsule manufactured at Takeda Pharmaceutical Company Ltd. (Osaka, Japan) (TPC).

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. This study will compare bioavailability of dexlansoprazole from 30 mg and 60 mg dexlansoprazole delayed release capsules manufactured at TOB relative to the corresponding 30 mg and 60 mg dexlansoprazole delayed release capsules manufactured at TPC. The study will enroll approximately 104 participants. Participants will be randomly assigned (by chance, like flipping a coin) to 1 of the 4 treatment sequences:

* Dexlansoprazole 30 mg TOB followed by Dexlansoprazole 30 mg TPC
* Dexlansoprazole 30 mg TPC followed by Dexlansoprazole 30 mg TOB
* Dexlansoprazole 60 mg TOB followed by Dexlansoprazole 60 mg TPC
* Dexlansoprazole 60 mg TPC followed by Dexlansoprazole 60 mg TOB

All participants will be asked to take single oral dose of dexlansoprazole at the same time on Day 1 of each Period. This single center trial will be conducted in the United States. The overall time to participate in this study is 18 days. Participants will visit the clinic on Day -1 and remained confined until Day 2 of Period 1 and 2. A washout period of minimum 5 days will be maintained between the doses in each Period. Participants will be contacted by telephone 10 (+/-2) days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women aged 18 to 55 years old, inclusive, with a body mass index between 18 and 30 kilogram per square meter (kg/m^2), inclusive.
2. Who are capable of understanding and complying with protocol requirements.
3. Must be in good health as determined by a physician based upon medical history, vital signs, electrocardiogram (ECG), and physical examination.
4. Must have clinical chemistry, hematology, and complete urinalysis (after fasting for at least 8 hours) at Screening and Check-in (Day -1 of Period 1) results within the reference range for the testing laboratory unless the out-of-range results are deemed not clinically significant by the investigator.
5. Must sign a written informed consent form (ICF) prior to initiation of study procedures.

Exclusion Criteria:

1. Has a history of significant gastrointestinal (GI) disorders manifested with persistent, chronic or intermittent nausea, vomiting, diarrhea, or has a current or recent (within 6 months) GI disease that would influence the absorption of drugs (example, a history of malabsorption, severe esophageal reflux, peptic ulcer disease or erosive esophagitis (EE) with frequent [more than once per week] occurrence of heartburn).
2. Has consumed medications, certain foods, and supplements, including prescription and over-the-counter medications, within the protocol-specified time periods prior to Check-in (Day -1 of Period 1), or is unwilling to agree to abstain from these products.
3. Have received dexlansoprazole in a previous clinical study or as a therapeutic agent within 6 months of Screening,
4. Have a known hypersensitivity to any component of the formulation of dexlansoprazole capsules or other drugs with the same mechanism of action (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole), or related compounds.
5. Any significant results from physical examination or clinical laboratory results that make the participant unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- PRAHS Phase 1 unit, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 25 April 2017 to 31 July 2017.
Pre-assignment Details: Healthy participants were enrolled in this 2 part study to receive dexlansoprazole 30 milligram (mg) capsules manufactured by Takeda GmbH Plant (Oranienburg, Germany) (TOB) or 30 mg capsules manufactured by Takeda Pharmaceutical Company Ltd. (Osaka, Japan) (TPC) in Part 1 and dexlansoprazole 60 mg capsules by TOB or 60 mg capsules by TPC in Part 2.
Groups:
- Part 1: Dexlansoprazole 30 mg TOB+ Dexlansoprazole 30 mg TPC: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (test), orally, once on Day 1 of Intervention Period 1 following a 10-hour fast, followed by minimum of 5-day washout period, further followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (reference) orally, once on Day 1 of Intervention Period 1 following a 10-hour fast.
- Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (reference), orally, once on Day 1 of Intervention Period 1 following a 10-hour fast, followed by minimum of 5-day washout period, further followed by dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (test) orally, once on Day 1 of Intervention Period 1 following a 10-hour fast.
- Part 2: Dexlansoprazole 60 mg TOB+ Dexlansoprazole 60 mg TPC: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (test), orally, once on Day 1 of Intervention Period 1 following a 10-hour fast, followed by minimum of 5-day washout period, further followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (reference) orally, once on Day 1 of Intervention Period 1 following a 10-hour fast.
- Part 2: Dexlansoprazole 60 mg TPC+ Dexlansoprazole 60 mg TOB: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (reference), orally, once on Day 1 of Intervention Period 1 following a 10-hour fast, followed by minimum of 5-day washout period, further followed by dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (test) orally, once on Day 1 of Intervention Period 1 following a 10-hour fast.
Period: Intervention Period 1 (2 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB+ Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB+ Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC+ Dexlansoprazole 60 mg TOB
Started | 28 | 28 | 30 | 30
Completed | 28 | 28 | 30 | 30
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (at Least 5 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB+ Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB+ Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC+ Dexlansoprazole 60 mg TOB
Started | 28 | 28 | 30 | 30
Completed | 27 | 23 | 26 | 25
Not Completed | 1 | 5 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1
Not completed — Other | 0 | 0 | 2 | 0
Period: Intervention Period 2 (2 Days)
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB+ Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB+ Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC+ Dexlansoprazole 60 mg TOB
Started | 27 | 23 | 26 | 25
Completed | 26 | 22 | 26 | 25
Not Completed | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dexlansoprazole 30 mg TOB+ Dexlansoprazole 30 mg TPC | Part 1: Dexlansoprazole 30 mg TPC + Dexlansoprazole 30 mg TOB | Part 2: Dexlansoprazole 60 mg TOB+ Dexlansoprazole 60 mg TPC | Part 2: Dexlansoprazole 60 mg TPC+ Dexlansoprazole 60 mg TOB | Total
Number analyzed (Participants) | 28 | 28 | 30 | 30 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.0 (7.95) | 28.5 (9.98) | 29.2 (7.78) | 28.4 (9.71) | 29.0 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 14 | 14 | 49
  Male | 17 | 18 | 16 | 16 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 1 | 17
  Not Hispanic or Latino | 21 | 22 | 25 | 29 | 97
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2 | 4
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  White | 26 | 24 | 28 | 25 | 103
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 30 | 30 | 116
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.7 (2.59) | 24.4 (2.75) | 24.6 (2.65) | 24.5 (3.33) | 24.5 (2.82)
Smoking Classification [Number; unit: participants]
  Never Smoked | 24 | 28 | 27 | 28 | 107
  Former Smoker | 4 | 0 | 3 | 2 | 9
  Current Smoker | 0 | 0 | 0 | 0 | 0
Alcohol Classification [Number; unit: participants]
  Never Drank | 19 | 19 | 18 | 18 | 74
  Former Drinker | 4 | 3 | 4 | 1 | 12
  Current Drinker | 5 | 6 | 8 | 11 | 30
Caffeine Consumption [Number; unit: participants]
  Had caffeine consumption | 15 | 15 | 18 | 22 | 70
  Had no caffeine consumption | 13 | 13 | 12 | 8 | 46
Xanthine Consumption [Number; unit: participants]
  Had xanthine consumption | 15 | 15 | 18 | 22 | 70
  Had no xanthine consumption | 13 | 13 | 12 | 8 | 46

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Dexlansoprazole
Time Frame: Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Groups:
- Dexlansoprazole 30 mg TOB: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TOB (test), orally, once on Day 1 of Intervention Period 1 or 2.
- Dexlansoprazole 30 mg TPC: Dexlansoprazole 30 mg, delayed-release capsule manufactured by TPC (reference), orally, once on Day 1 of Intervention Period 1 or 2.
- Dexlansoprazole 60 mg TOB: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TOB (test), orally, once on Day 1 of Intervention Period 1 or 2.
- Dexlansoprazole 60 mg TPC: Dexlansoprazole 60 mg, delayed-release capsule manufactured by TPC (reference), orally, once on Day 1 of Intervention Period 1 or 2.
Arm/Group | Dexlansoprazole 30 mg TOB | Dexlansoprazole 30 mg TPC | Dexlansoprazole 60 mg TOB | Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 51 | 55 | 55 | 56
nanogram/milliliter (ng/mL) | 515.7 (257.60) | 519.5 (305.66) | 1027.0 (598.74) | 978.6 (581.34)
Statistical Analysis 1: Comparison: Dexlansoprazole 30 mg TOB vs Dexlansoprazole 30 mg TPC; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with regimen, sequence and period as a fixed effect and subject nested within sequence as a random effect. The least squares means and difference of least squares means for the log-transformed parameters were exponentiated to obtain the point estimates and 90 percent (%) confidence intervals (CIs) on the original scale; p = 0.5535, ANOVA; Least square (LS) mean ratio = 1.0436, 90% CI 2-sided [0.9453 to 1.1521]
Statistical Analysis 2: Comparison: Dexlansoprazole 60 mg TOB vs Dexlansoprazole 60 mg TPC; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with regimen, sequence and period as a fixed effect and subject nested within sequence as a random effect. The least squares means and difference of least squares means for the log-transformed parameters were exponentiated to obtain the point estimates and 90% CIs on the original scale; p = 0.8920, ANOVA; LS mean ratio = 1.0185, 90% CI 2-sided [0.9334 to 1.1113]

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Dexlansoprazole
Time Frame: Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter(ng*hour/mL)
Arm/Group | Dexlansoprazole 30 mg TOB | Dexlansoprazole 30 mg TPC | Dexlansoprazole 60 mg TOB | Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 51 | 55 | 55 | 56
nanogram*hour per milliliter(ng*hour/mL) | 2416.3 (2280.91) | 2327.6 (2052.94) | 5715.5 (4521.84) | 5684.7 (5361.88)
Statistical Analysis 1: Comparison: Dexlansoprazole 30 mg TOB vs Dexlansoprazole 30 mg TPC; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.3209, ANOVA; LS mean ratio = 1.0390, 90% CI 2-sided [0.9792 to 1.1024]
Statistical Analysis 2: Comparison: Dexlansoprazole 60 mg TOB vs Dexlansoprazole 60 mg TPC; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.3896, ANOVA; LS mean ratio = 1.0353, 90% CI 2-sided [0.9719 to 1.1029]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Dexlansoprazole
Time Frame: Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose
Population: The PK set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration. PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Dexlansoprazole 30 mg TOB | Dexlansoprazole 30 mg TPC | Dexlansoprazole 60 mg TOB | Dexlansoprazole 60 mg TPC
Number analyzed (Participants) | 51 | 55 | 55 | 56
ng*hour/mL | 2579.6 (2760.38) | 2420.6 (2322.58) | 5746.2 (4785.72) | 5630.4 (5527.34)
Statistical Analysis 1: Comparison: Dexlansoprazole 30 mg TOB vs Dexlansoprazole 30 mg TPC; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.4163, ANOVA; LS mean ratio = 1.0335, 90% CI 2-sided [0.9733 to 1.0975]
Statistical Analysis 2: Comparison: Dexlansoprazole 60 mg TOB vs Dexlansoprazole 60 mg TPC; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.9778, ANOVA; LS mean ratio = 1.0031, 90% CI 2-sided [0.9458 to 1.0638]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Day 37)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole 30 mg TOB | Dexlansoprazole 30 mg TPC | Dexlansoprazole 60 mg TOB | Dexlansoprazole 60 mg TPC
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/55 | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/55 | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 8/51 | 9/55 | 8/55 | 11/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 30 mg TOB (N=51) | Dexlansoprazole 30 mg TPC (N=55) | Dexlansoprazole 60 mg TOB (N=55) | Dexlansoprazole 60 mg TPC (N=56)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site erosion (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT03131895/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03131895/SAP_001.pdf